CLINICAL TRIAL: NCT05553977
Title: Design and Validation of an Artificial Intelligence System to Detect the Quality of Colon Cleansing Before Colonoscopy
Brief Title: Artificial Intelligence and Bowel Cleansing Quality
Acronym: CALPER2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Other Study IDs: CNN bowel cleansing
Record Dates: First submitted 2022-09-19; First posted 2022-09-26 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Cleansing Quality of the Colon
Keywords: Bowel cleansing; Colonoscopy; Convolutional Neural Network
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive patients for outpatient colonoscopy: The researchers will offer to participate in the study to patients scheduled for a colonoscopy who meet all the inclusion criteria and none of the exclusion criteria
  Interventions: Drug: Bowel preparation for colonoscopy; Procedure: Colonoscopy

INTERVENTIONS:
Drug: Bowel preparation for colonoscopy — one day liquid diet will be administered to every patient included in the study and: split-dose bowel preparation with 4 Liters of Polyethylene glycol solution, 2 Liters of PEG-Ascorbic acid or 2 Liters Picosulfate.
Procedure: Colonoscopy — Colonoscopy will be performed to every patient included in the study

SUMMARY:
The main purpose of the study is to design and validate a convolutional neural network (CNN) with the ability to discriminate between pictures of effluents with different qualities of bowel cleansing and in a second time to prospectively assess in a cohort of patients the agreement between the result of the last rectal effluent quality assessed by the CNN and the cleansing quality assessed during the colonoscopy assessed by a validated scale (Boston Bowel Preparation Scale, BBPS). Patients will be prepared with polyethylene glycol (PEG), PEG plus ascorbic acid (PEG-Asc) or sodium picosulfate-oxide magnesium solution (PS).

DETAILED DESCRIPTION:
The patient perception of the last bowel movement before the colonoscopy has been shown a powerful predictor of bowel cleansing rated during colonoscopy. A large study involving 1011 patients distributed in a derivation cohort (633 patients) and a validation cohort (378 patients) using a set of 4 pictures resembling bowel cleansing qualities showed a moderate agreement with the BBPS. In addition, a good agreement was found when the staff perception and patient perception of the last bowel movement were compared. These findings offer an excellent opportunity to test rescue cleansing interventions the same day of the examination, before colonoscopy.

Over the last two years, artificial intelligence applications have wrought a substantial breakthrough in several disciplines, including endoscopy. Machine learning and its more advanced form deep learning, refers to the development of algorithms (convolutional neural networks) with the ability to learn and perform certain tasks. In the endoscopy setting, computer vision applications have been stated as research priority field. Based on all this experience, the aim of this study was to design and to validate a convolutional neural network capable of automatically predicting the quality of the patient cleansing at home after the intake of the bowel cleansing solution and before attending the colonoscopy. The other aim was to prospectively assess in a cohort of patients the agreement between the result of the last rectal effluent quality assessed by the convolutional neural network and the cleansing quality assessed during the colonoscopy assessed by a validated scale (Boston Bowel Preparation Scale, BBPS) This study is nested in an observational prospective study conducted at the Open Access Endoscopy Unit of the Hospital Universitario de Canarias between February 2021 and May 2021 (NCT04702646). A total of 633 consecutive outpatients with a scheduled colonoscopy participated in this study (a total of 266 patients (42%) sent at least one picture). After this study, patients in whom an outpatient colonoscopy was requested, were asked to provide pictures of their effluents during bowel preparation intake. A subgroup of these images will be classified by the personal of our unit in adequate and inadequate and will be used to train the convolutional neural network. Another set of images will be used to validate the convolutional neural network. Additionally, the investigators will validate in-vivo the convolutional neural network comparing its classification of the effluent quality with a validated colon cleansing scale during the colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age >18, to sign the informed consent,
* Patients with indication of outpatient colonoscopy
* Patients ingesting the bowel preparation

Exclusion Criteria:

* Incomplete colonoscopy (except for poor bowel preparation)
* Contraindication for colonoscopy
* Allergies.
* Refusal to participate in the study or impairment to sign the informed consent.
* Colectomy (more than 1 segment)
* Dementia with difficulty in the intake of the preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The researchers will offer to participate in the study to patients scheduled for a colonoscopy who meet all the inclusion criteria and none of the exclusion criteria. The researchers will explain the purpose of the study and will ask to sign the informed consent. They will give verbal and written information.
Sampling Method: Non-Probability Sample
Enrollment: 667 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Effluent characteristics | 1 year
  Effluent characteristics. Set of 4 pictures categorized in adequate preparation (clear liquid, clear liquid with lumps) and inadequate preparation (dark liquid, or dark liquid with solid particles). The concolutional Neural Network will be trained with effluent images and validated.
Quality of bowel cleansing assessed by the Boston Bowel Preparation Scale | 1 years
  Quality of bowel cleansing assessed by the Boston Bowel Preparation Scale. This scale goes from 0 (no preparation) to 3 points (excellent preparation) in the three segments of the colon (proximal, transverse and distal). The maximum score is 9 points

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, San Cristóbal de La Laguna, S/C de Tenerife, Spain

REFERENCES:
- [Result] Mori Y, Misawa M, Kudo SE. Challenges in artificial intelligence for polyp detection. Dig Endosc. 2022 May;34(4):870-871. doi: 10.1111/den.14279. Epub 2022 Mar 22. No abstract available. PMID 35318734
- [Result] Berzin TM, Parasa S, Wallace MB, Gross SA, Repici A, Sharma P. Position statement on priorities for artificial intelligence in GI endoscopy: a report by the ASGE Task Force. Gastrointest Endosc. 2020 Oct;92(4):951-959. doi: 10.1016/j.gie.2020.06.035. Epub 2020 Jun 19. PMID 32565188
- [Result] Fatima H, Johnson CS, Rex DK. Patients' description of rectal effluent and quality of bowel preparation at colonoscopy. Gastrointest Endosc. 2010 Jun;71(7):1244-1252.e2. doi: 10.1016/j.gie.2009.11.053. Epub 2010 Apr 1. PMID 20362286
- [Result] Alzubaidi L, Zhang J, Humaidi AJ, Al-Dujaili A, Duan Y, Al-Shamma O, Santamaria J, Fadhel MA, Al-Amidie M, Farhan L. Review of deep learning: concepts, CNN architectures, challenges, applications, future directions. J Big Data. 2021;8(1):53. doi: 10.1186/s40537-021-00444-8. Epub 2021 Mar 31. PMID 33816053
- [Result] Harewood GC, Wright CA, Baron TH. Assessment of patients' perceptions of bowel preparation quality at colonoscopy. Am J Gastroenterol. 2004 May;99(5):839-43. doi: 10.1111/j.1572-0241.2004.04176.x. PMID 15128347